CLINICAL TRIAL: NCT06809933
Title: EMPOWER: Exercise and Movement to Promote Our Patients With (Gynecologic) Cancer to Enhance Resiliency
Brief Title: Exercise and Movement to Enhance Resiliency in Cancer Patients
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Sword Health, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 244013; NCI-2025-00773 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Cancer
Keywords: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Digital Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1: EMPOWER Feasibility Cohort (Experimental): The first 20 participants enrolled with receive the EMPOWER intervention which consists of the "Move" mobile application that synchronizes with a FitBit that tracks heart rate, step count, and motion and also receive UCSF-based, online peer support network with individual and small group sessions that occur every four weeks. Questionnaires will be given at baseline, week 9, the end of treatment, and at 3 months after completion of the interventions.
  Interventions: Other: Digital Health Mobile App; Other: Virtual Support Group; Other: Health Coaching
- Stage 2: EMPOWER (Experimental): Participants randomized to the EMPOWER intervention will receive the "Move" mobile application that synchronizes with a FitBit that tracks heart rate, step count, and motion and also receive UCSF-based, online peer support network with individual and small group sessions that occur every four weeks. Questionnaires will be given at baseline, week 9, the end of treatment, and at 3 months after completion of the interventions.
  Interventions: Other: Digital Health Mobile App; Other: Virtual Support Group; Other: Health Coaching
- Stage 2: Enhanced usual care (EUS) (Active Comparator): Participants randomized to the EUS group will receive a similar kit that includes a FitBit (equivalent features to what the intervention arm receives), and receive a handout that details recommended national guidelines on exercise during cancer treatment. Participants will be asked to allow the FitBit to be linked to a study email that provides a summary of weekly activity to track activity throughout the study.
  Interventions: Other: FitBit; Other: Handouts

INTERVENTIONS:
Other: Digital Health Mobile App — A digital health technology (DHT) called "Move" by Sword Health, which utilizes a mobile app displaying tailored and recommended exercise options, wearable technology (Move wearable or equivalent), and a web-based platform monitored by a physical therapist who will provide individual support
  Other Names: Digital health technology (DHT); Move App
  Arms: Stage 1: EMPOWER Feasibility Cohort; Stage 2: EMPOWER
Other: Virtual Support Group — An institutional, virtual peer support group session will include a maximum of 5 participant per group
  Other Names: Video Support Group
  Arms: Stage 1: EMPOWER Feasibility Cohort; Stage 2: EMPOWER
Other: Health Coaching — The facilitated group and discussions sessions will be led by a University of California, San Francisco (UCSF) certified health coach (CHC), following a pre-specified agenda and provided virtually
  Other Names: Virtual Health Coach; Certified Health Coach
  Arms: Stage 1: EMPOWER Feasibility Cohort; Stage 2: EMPOWER
Other: FitBit — FitBit is a health and activity tracking device placed around the wrist
  Other Names: Activity Tracking Device
  Arms: Stage 2: Enhanced usual care (EUS)
Other: Handouts — A handout with exercise recommendations for those with cancer in accordance with national guidelines
  Other Names: Study Handouts
  Arms: Stage 2: Enhanced usual care (EUS)

SUMMARY:
This is a single-center, pilot, hybrid type 1 design implementation study to evaluate the feasibility and implementation of a personalized digital exercise program and a virtual support group to improve patient-centered outcomes in patients receiving treatment for gynecologic cancer receiving treatment at University of California, San Francisco.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Stage 1 (single-arm pilot of intervention)

I. To assess the feasibility of recruitment of the EMPOWER intervention.

II. To assess the acceptability of the Exercise and Movement to Enhance Resiliency in Cancer Patients (EMPOWER) intervention.

Stage 2 (pilot randomized study comparing EMPOWER to enhanced usual care (EUS).

I. To assess the feasibility of recruitment of the study when randomized.

II. To assess the acceptability of a randomized study (in both groups)

SECONDARY OBJECTIVES:

Stage 1 and 2

I. To evaluate retention and adherence of the interventions.

II. To evaluate the components of acceptability and adherence of the interventions.

III. To evaluate changes in objective physical activity measures as a single arm pilot study (stage 1) and compared to EUS (stage 2) of the EMPOWER intervention.

IV. To evaluate changes in improving patient reported quality of life measures as a single arm pilot study (stage 1) and compared to EUS (stage 2) of the EMPOWER intervention.

OUTLINE:

Participants will be enrolled in 2 stages.

Stage 1 is a single-arm pilot study testing the EMPOWER intervention to gather feedback for refinement and optimization of the program to implement in Stage 2.

Stage 2 is a pilot, randomized trial where participants will be assigned in a 1 to 1 ratio to either the EMPOWER program or EUS. All participants will be stratified by treatment type (neoadjuvant versus adjuvant therapy).

Participants will be enrolled in these interventions for a total of 16 weeks and receive a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Newly diagnosed with a gynecological cancer (including ovarian tubal or peritoneal, uterine, cervical, vaginal, vulvar, and/or gestational trophoblastic neoplasia) and currently undergoing treatment chemotherapy, surgery, etc.).
3. Able to understand study procedures and to comply with study procedures for the entire length of the study.
4. Ability to understand a written informed consent document, and the willingness to sign it.
5. Eastern Cooperative Oncology Group (ECOG) status < 4.
6. Willingness to participate and wear an activity tracker (FitBit).
7. Planning to start systemic treatment or currently receiving Cycle 1 of systemic treatment.

Exclusion Criteria:

1. Medically ineligible or contraindications to exercise as determined by their oncologist; or contradiction to any other study-related procedure or assessment.
2. Cognitive or visual impairments that would limit participant's ability to utilize and interact with the DHT platform. Note: If a visually impaired participant has a caregiver who can help them use the DHT platform, the participant will not be excluded.
3. Existing performance of excessive physical activity (>210 minutes per week of moderate to vigorous intensity exercise at baseline).
4. Existing enrollment in an exercise program or physical therapy program.
5. Inability to speak and read English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2031-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (Stage 1) | Up to 20 days
  Feasibility of the intervention is defined as >= 30% recruitment rate for participants in Stage 1.
Recruitment Rate (Stage 2) | Up to 20 days
  Feasibility of the intervention is defined as >= 30% recruitment rate for participants in Stage 2.
Enrollment Rate (Stage 1) | Up to 20 days
  Feasibility of the intervention is defined as > 30% enrollment rate for participants in Stage 1.
Enrollment Rate (Stage 2) | Up to 20 days
  Feasibility of the intervention is defined as > 30% enrollment rate for participants in Stage 2.
Percentage of participants recommending the EMPOWER intervention (Stage 1 & 2, EMPOWER Participants only) | 1 day
  Acceptability of the intervention will be measured by a physician designed questionnaire assessing the acceptability of the EMPOWER intervention. The questionnaire is an 8-item measure of which assesses participants perceived acceptability of the EMPOWER program. Each item response falls on a scale of 1 (Strongly disagree) to 5 (Strongly agree). The percentage of participants with a response of either agree or strongly agree will be reported.
Percentage of participants adherence to the intervention (Stage 2, EMPOWER Participants only) | Up to 16 weeks
  Adherence to the intervention will be measured for each participant, from week 1 to study completion per data collected by wearable device and by CHC collection. The percentage of participants will be reported

SECONDARY OUTCOMES:
Retention Rate | Up to 16 weeks
  The retention rate of participants in both groups will be reported as a percentage of participants. Retention is defined as >50% of the participants
Percentage of participants who completed prescribed exercises | Up to 16 weeks
  The percentage of participants who completed at least 50% of prescribed exercises will be reported
Percentage of participants who utilized the mobile application | Up to 16 weeks
  The percentage of participants who utilized at least 75% of the mobile application will be reported.
Percent attendance of the online meetings | Up to 16 weeks
  The percentage of participants who attended at least 50% of the online peer support sessions will be reported
Mean changes in average step count over time | Up to 16 weeks
  The mean change in average step count as measured by the wearable device (Move wearable or equivalent) and actigraphy for participants as tracked by a wearable device will be reported along with a 90% confidence interval
Mean changes in the minutes participants were active over time | Up to 16 weeks
  The mean change in average active time as measured in minutes by the wearable device will be reported along with a 90% confidence interval
Mean changes in scores on the short performance physical battery (SPPB) survey over time | Up to 16 weeks
  The SPPB is an objective measurement instrument developed by the National Institute of Aging (NIA) to measure balance, lower extremity strength, and functional capacity in older adults (>65 years of age). The test includes three different domains (walking, sit-to-stand and balance activities and are assessed and assigned points by a physician or study staff to assess overall functional mobility. Each task is assigned a number of points or a confirmation of completion, with higher points or task completion indicating better balance, better extremity strength, and higher functional capacity. will be performed via video visit. Each component is scored from 0-4 with a total of 12 with higher scores predictive of immobility, reduced activities of daily living (ADLs), and falls.
Mean changes in scores on the Patient Reported Outcomes Measurement Information System-Cancer (PROMIS) Global Health v1.2 | Up to 7 months
  The Patient Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 - Global Health (also referred to as PROMIS-10) is a ten-item patient reported measure of physical, mental and social health. Items query general health, quality of life, physical health, mental health, satisfaction with discretionary social activities, carrying out every day physical activities, pain, fatigue, satisfaction with social roles, and emotional problems. with a response ranging from 1="Poor" to 5="Excellent" with 1 item addressing pain with a raw score range of 0 "No pain at all" to 10="Worst possible pain". The total raw score ranging from 4 - 50, which are converted to a scaled T-score (range of 16.2 - 67.7) with higher scores indicating a greater overall quality of life. Mean changes in the global score will be reported along with a 90% confidence interval.
Mean changes in scores on Patient Reported Outcomes Measurement Information System-Cancer (PROMIS) Physical function (PF) 10b | Up to 7 months
  The PROMIS PF 10b is a 10-item questionnaire which measures respondents' self-reported capability to physically function in the context of cancer and/or cancer treatment experiences with a response ranging from 1="Not at all" to 5="Cannot do", and a total raw score ranging from 10 - 50, which are converted to a scaled T-score (range of 13.8 - 61.3) with higher scores indicating a greater hinderance to engagement in physical activities. The mean change in scores along with a 90% confidence interval will be reported.
Mean changes in scores on the Patient Reported Outcomes Measurement Information System-Cancer (PROMIS) Fatigue- Short Form 4a | Up to 7 months
  This 4-item questionnaire to measure fatigue based on responses to statements about how the participants feel with a response ranging from 1="Not at all" to 5="Very Much", and a total raw score ranging from 4 - 20, which are converted to a scaled T-score (range 33.7 to 75.8) with higher scores indicating a greater feeling of fatigue. The mean change in scores along with a 90% confidence interval will be reported.
Mean changes in scores on the Generalized Anxiety Disorder Questionnaire (GAD-7) over time | Up to 7 months
  The GAD-7 is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater. The mean change in scores along with a 90% confidence interval will be reported.
Mean changes in scores on the Life Space Assessment (LSA) | Up to 7 months
  The LSA is a 5-item questionnaire assessing mobility in adults. Each item on the assessment is associated with 3 factors: Accessing Spaces (0=No, 1=Yes), Frequency (1=Less than 1/week up to 4=Daily), and Independence (1=Personal assistance needed to 2=No equipment or personal assistance needed). Each space level is scored by Accessing Spaces score x Frequency score x Independence score. The total LSA score is calculated by taking the sum of each of the 5 items. Higher scores indicate a higher usage of life space.
Mean changes in scores on the Functional Assessment of Cancer Therapy (FACT)/Gynecologic Oncology Group (GOG) - Neurotoxicity (FACT/GOG-NTX) | Up to 7 months
  The FACT/GOG-NTX is a 38-item questionnaire to assess symptoms quality of life and peripheral neuropathy in cancer patients undergoing chemotherapy. The FACT/GOG-NTX item responses range from 0 (not at all) to 4 (very much). To calculate the FACT/GOG-Ntx Trial Outcome Index (TOI) score, the sum of the item scores from the physical well-being subscale, the functional well-being subscale and the neurotoxicity subscale are combined to create a TOI score ranging from 0-100 with higher scores indicating a better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cham, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No